CLINICAL TRIAL: NCT06465537
Title: A Clinical Study on CRISPR/Cas9 Instantaneous Gene Editing Therapy to Primary Open-angle Glaucoma With Elevated Intraocular Pressure and MYOC Gene Mutation
Brief Title: CRISPR/Cas9 Instantaneous Gene Editing Therapy to Intraocular Hypertensive POAG With MYOC Mutation
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Shanghai BDgene Co., Ltd. (Industry)
Collaborators: Beijing Tongren Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: BD-MMG-113001
Record Dates: First submitted 2024-06-13; First posted 2024-06-20 (Actual); Last update posted 2024-06-24 (Actual); Status verified 2024-06

CONDITIONS: Primary Open Angle Glaucoma
Keywords: primary open angle glaucoma; POAG; elevated intraocular pressure; MYOC gene mutation
MeSH Terms: conditions — Glaucoma, Open-Angle; Ocular Hypertension

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1: POAG without vision for interventional eye (Experimental): Interventional eye of participants with POAG has no vision, with mutated or unmutated MYOC gene. Single dose of BD113vVLP will be administrated intracamerally for target interventional eye.
  Interventions: Genetic: BD113vVLP
- Group 2: POAG with vision for interventional eye (Experimental): Interventional eye of participants with POAG has vision acuity, and MYOC gene mutation test is positive. Single dose of BD113vVLP will be administrated intracamerally for target interventional eye.
  Interventions: Genetic: BD113vVLP

INTERVENTIONS:
Genetic: BD113vVLP — CRISPR/Cas9 gene editing technology, called BD113vVLP (also BD113 virus-like particle) which is a developing product of gene therapy from modified third-generation integrated defective lentivirus, can deliver gRNA/Cas9 ribonucleoprotein complex (RNP). It works to knock out or knock down the mutated MYOC gene. The BD113vVLP is administrated by intracamerally injecton (sigle-dose: 4ug/p24) for each target interventional eye.
  Other Names: BD113 virus-like particle; CRISPR/Cas9 mRNA instantaneous gene editing technology

SUMMARY:
This study is intented to evaluate the safety, tolerability and preliminary efficacy of CRISPR/Cas9 Instantaneous Gene Editing Therapy (BD113 virus-like particle, also BD113vLVP) in patients with primary open-angle glaucoma (POAG) with elevated intraocular pressure and MYOC gene mutation. The main objectives to evaluate the safety and tolerability BD113vLVP) in POAG patients with intraocular hypertension and MYOC mutation, and secondary objectives is to explore the preliminary efficacy and the metabolism characteristics of BD113vLVP in participants.

DETAILED DESCRIPTION:
This is an open, single-dose, two-arm, non-randomised clinical study. A total of 6 to 9 POAG patients with high intraocular pressure were enrolled and divided into two test groups. Test Group 1 recruits 3 POAG patients, who have elevated IOP and positive or negative MYOC mutation and target interventing eye is no vision. Test Group 2 will recruit 3 to 6 POAG patients with MYOC mutations and visual acuity. In order to better verify the lowering IOP effectiveness of BD113vVLP, another 2 or 3 participants will be recruied in Group 2 on-demand. Each participant will receive single dosing BD113vVLP (4µg p24) by intracameral injection in the interventing eye, then conduct the evaluations of the safety and efficacy according to visit schedule in 1 year follow-up。

ELIGIBILITY:
Inclusion Criteria:

1. Signed ICF;
2. Aged 18 to 65 years old;
3. Primary open Angle glaucoma (POAG) with elevated intraocular pressure (IOP) was diagnosed with ≥1 year medical history record ;
4. Good function level of organs;
5. Good compliance and willing to comply with the visit schedule, laboratory tests and other specified test etc. per protocol;
6. Agreeing to accept a long-term safety follow-up after 1 year of study.

Special Inclusion Criteria for Group 1:

* Target intervenning eye is no visual acuity;
* The intraocular pressure (IOP) was ≤35 mmHg and > 21 mmHg after receiving a combination therapy of 2 or more drugs lowering IOP.

Special Inclusion Criteria for Group 2:

* MYOC gene mutation was detected in peripheral blood nucleated cells ;
* The intraocular pressure (IOP) was ≤30 mmHg and > 21 mmHg after receiving a combination therapy of 2 or more drugs lowering IOP;
* Both eyes have a Shaffer Angle mirror rating greater than 3.

Exclusion Criteria:

1. Secondary glaucoma;
2. Any active or recurrent intraocular infection or inflammation, including but not limited to uveitis;
3. The target intervenning eye has severe xerophthalmia or clinically significant active corneal disease;
4. Any condition no accepting the measure of IOP;
5. Any positive of human immunodeficiency virus type 1/2 (HIV-1/HIV-2) antibody, treponema pallidum (TP) specific antibody, human T-lymphotropic virus type 1 or 2 (HTLV-1/HTLV-2) antibody, or vesicular stomatitis virus G (VSV-G) antibody;
6. Any of hepatitis B virus (HBV) HbsAg or HBV-DNA, hepatitis C virus (HCV) HCAb, or epstein-barr virus (EBV), or cytomegalovirus (CMV) nucleic acid test is positive;
7. Severe active bacterial, viral, fungal, malaria or parasitic systemic infection;
8. Any past or present malignancy, myeloproliferative or immunodeficient disease;
9. History of major organ diseases or abnormalities in laboratory tests, including:

   1. Liver cirrhosis, liver fibrosis or active hepatitis, and/or abnormal liver function tests (serum total bilirubin (TBIL) ≥1.5 x upper limit of normal (ULN); Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≥2.5×ULN; Alkaline phosphatase ≥2.5 × ULN);
   2. Cardiovascular and cerebrovascular diseases, including uncontrolled hypertension, myocardial infarction, myocarditis, arrhythmia, stroke, etc.;
   3. Kidney disease, or creatinine ≥ 1.5ULN and creatinine clearance < 30% normal level (using the Cockcroft-Gault equation);
   4. Endocrine disorders, such as insulin-dependent diabetes mellitus, hyperthyroidism or hypothyroidism;
   5. Severe pulmonary hypertension, chronic obstructive pulmonary disease, interstitial pneumonia;
10. Any severe psychiatric disorders;
11. Participating in another clinical study of a drug or device, or administrated the investigational drug within 42 days prior to the screening visit;
12. Pregnant or lactating women;
13. Refusing to accept any contraception measures;
14. Allergic to clinical investigational drugs or their excipients;
15. Other conditions assessed by the investigator as unsuitable for participation in this study.

Special Exclusion Criteria for Group 2:

* Retinal diseases: complicated with unexplained quadrant blindness, neovascularization age-related macular degeneration, retinal branch vein obstruction, central retinal vein obstruction, cystoid macular edema, macular hiatal hole and central serous retinopathy;
* A history of anterior chamber angle stenosis, congenital glaucoma, or angle closure, clinically significant anterior peripheral adhesion, or extensive cicatricial adhesion caused by surgery/laser therapy in the anterior chamber angle;
* The central corneal thickness is less than 480 μm or more than 620 μm.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Estimated)
Dates: Start 2024-06-10 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Ocular adverse events (AEs) | 12 months
  The charactaristics of ocular adverse events include endophthalmitis, hypopyon, hyphaema and corneal injection site reaction etc. will be evaluated at Week 1, Week 2, Week 3, Week 4, Month 6 and Month 12 after BD113vVLP administration.
Number and percentage of participants whose IOP decrease ≤21 mmHg | 12 months
  at Month 1, Month 2, Month 3, Month 6 and Month 12 after BD113vVLP administration

SECONDARY OUTCOMES:
Systemic adverse events (AEs): The type, number and incidence of AEs and serious adverse events (SAEs) | 12 months
  Systemic adverse events (AEs): The type, number and incidence of AEs and serious adverse events (SAEs) will be analysized within 12 months after BD113vVLP administration.
Number and percentage of participants whose IOP decrease by ≥ 20% from baseline | 12 months
  at Month 1, Month 2, Month 3, Month 6 and Month 12 after BD113vVLP administration
Any ocular maligancies related to BD113vVLP | 12 months
  after BD113vVLP administration
Changes in BCVA from baseline | 12 months
  at Month 3, Month 6 and Month 12 after BD113 vVLP administration, not applicable to group 1.
Changes in visual fields from baseline | 12 months
  at Month 3, Month 6 and Month 12 after BD113 vVLP administration, not applicable to group 1.
Changes in RNFL from baseline | 12 months
  at Month 3, Month 6 and Month 12 after BD113 vVLP administration, not applicable to group 1.
P24 and Cas9 proteins concentration in aqueous humor | 1 months
  at hour 0 and Month 1 after BD113vVLP administration
P24 and Cas9 proteins concentration in blood | 7 days
  at hour 0 and Day 7 after BD113vVLP administration
Blood antibodies of anti-p24 protein and anti-Cas9 proteins | 12 months
  at Month 6 and Month 12 after BD113vVLP administration

CONTACTS AND LOCATIONS:
Overall Officials: Yufei Teng, M.D., Study Director — Beijing Tongren Hospital
Locations (1):
- Beijing Tongren Hospital, Capital Medical University, Beijing, Beijing Municipality, China